CLINICAL TRIAL: NCT02480764
Title: A Phase 3, Double-Blind, Randomized, Parallel-Group Study to Compare the Efficacy and Safety of TAK-491 With Valsartan in Chinese Subjects With Essential Hypertension
Brief Title: Azilsartan Medoxomil (TAK-491) Compared to Valsartan in Chinese Participants With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491_305; U1111-1159-5579 (Registry Identifier: WHO)
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Essential Hypertension
Keywords: Drug therapy
MeSH Terms: conditions — Essential Hypertension | interventions — azilsartan medoxomil; azilsartan; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan medoxomil 40 mg (Experimental): Run-in Period: azilsartan medoxomil 40 mg placebo-matching tablets, azilsartan medoxomil 80 mg placebo-matching tablets, and valsartan two 80 mg placebo-matching capsules, orally, once daily, for 2 weeks prior to the start of the treatment period. Treatment Period: azilsartan medoxomil 40 mg tablets, orally, once daily, azilsartan medoxomil 80 mg placebo-matching tablets, orally, once daily, and valsartan two 80 mg placebo-matching capsules, orally, once daily, for up to 8 weeks.
  Interventions: Drug: Azilsartan medoxomil; Drug: Azilsartan medoxomil Placebo; Drug: Valsartan Placebo
- Azilsartan medoxomil 80 mg (Experimental): Run-in Period: azilsartan medoxomil 40 mg placebo-matching tablets, azilsartan medoxomil 80 mg placebo-matching tablets, and valsartan two 80 mg placebo-matching capsules, orally, once daily, for 2 weeks prior to the start of the treatment period. Treatment Period: azilsartan medoxomil 80 mg tablets, orally, once daily, azilsartan medoxomil 40 mg placebo-matching tablets, orally, once daily, and valsartan two 80 mg placebo-matching capsules, orally, once daily, for up to 8 weeks.
  Interventions: Drug: Azilsartan medoxomil; Drug: Azilsartan medoxomil Placebo; Drug: Valsartan Placebo
- Valsartan 160 mg (Active Comparator): Run-in Period: azilsartan medoxomil 40 mg placebo-matching tablets, azilsartan medoxomil 80 mg placebo-matching tablets, and valsartan two 80 mg placebo-matching capsules, orally, once daily, for 2 weeks prior to the start of the treatment period. Treatment Period: valsartan two 80 mg capsules, orally, once daily, azilsartan medoxomil 40 mg placebo-matching tablets, orally, once daily, and azilsartan medoxomil 80 mg placebo-matching tablets, orally, once daily, for up to 8 weeks.
  Interventions: Drug: Valsartan; Drug: Azilsartan medoxomil Placebo; Drug: Valsartan Placebo

INTERVENTIONS:
Drug: Azilsartan medoxomil — Azilsartan medoxomil tablets
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan medoxomil 40 mg; Azilsartan medoxomil 80 mg
Drug: Valsartan — Valsartan 80 mg capsules
  Other Names: Diovan®
  Arms: Valsartan 160 mg
Drug: Azilsartan medoxomil Placebo — Azilsartan medoxomil placebo-matching tablets
Drug: Valsartan Placebo — Valsartan placebo-matching capsules

SUMMARY:
The purpose of this study is to evaluate the antihypertensive effect of azilsartan medoxomil compared with valsartan in Chinese participants with essential hypertension.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-491 (azilsartan medoxomil). Azilsartan medoxomil is being tested to treat Chinese people who have essential hypertension. This study will look at change in blood pressure after 8 weeks of treatment in people who take azilsartan medoxomil compared to people who take valsartan.

The study enrolled 612 patients. Prior to the start of study treatment, participants who have not received antihypertensive treatment within 28 days participated in a 2-week -run in period. Upon completion of the run-in period, participants were randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* azilsartan medoxomil 40 mg
* azilsartan medoxomil 80 mg
* Valsartan 160 mg

All participants were asked to take study medication at the same time each day throughout the study.

This multi-centre trial was conducted in China. The overall time to participate in this study is up to 14 weeks. Participants made 9 visits to the clinic and contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is treated with antihypertensive therapy and has a post-washout mean sitting clinic systolic blood pressure (SBP) ≥150 and ≤180 mm Hg on Day 1; or the participant has not received antihypertensive treatment within 28 days prior to Screening and has a mean sitting clinic SBP ≥150 and ≤180 mm Hg at the Screening Visit and on Day 1.
2. Is a man or woman aged 18 years or older.
3. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
4. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
5. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent through 30 days after last study drug dose.
6. Has clinical laboratory test results (clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or the investigator does not consider the results to be clinically significant.
7. Is willing to discontinue current antihypertensive medications on Day -21 or on Day -28 if the participant is on amlodipine or chlorthalidone.

Exclusion Criteria:

1. Has a mean, sitting clinic diastolic blood pressure (DBP) greater than 110 mm Hg at Day 1 (after placebo run in).
2. Is non-compliant (less than 70% or greater than 130%) with study medication during placebo run-in period.
3. Has secondary hypertension of any etiology (eg, renovascular disease documented as the cause of hypertension, pheochromocytoma, Cushing's syndrome).
4. Has a history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
5. Has clinically significant cardiac conduction defects (eg, third-degree atrioventricular block, sick sinus syndrome).
6. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease and hypertrophic obstructive cardiomyopathy (HOCM).
7. Has severe renal dysfunction or disease (based on estimated glomerular filtration rate [GFR] <30 mL/min/1.73 m^2) at Screening.
8. Has known or suspected unilateral or bilateral renal artery stenosis.
9. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those participants with basal cell or Stage 1 squamous cell carcinoma of the skin).
10. Has type 1 or poorly controlled type 2 diabetes mellitus (hemoglobin A1c [HbA1c] >8.5%) at Screening.
11. Has hyperkalemia (defined as serum potassium above the normal reference range of the central laboratory) at Screening.
12. Has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level of greater than 2.5 times the upper limit of normal (ULN), active liver disease, or jaundice at Screening.
13. Has any other known serious disease or condition at Screening (or Randomization) that would compromise participant safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
14. Has a history of hypersensitivity or allergies to TAK-491 (azilsartan medoxomil), any of its excipients or other angiotension II (AII) receptor blockers (ARBs).
15. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
16. Is currently participating in another investigational study or is receiving or has received any investigational compound within 30 days prior to the first dose of study medication.

    Note: This criterion does not apply to participants who participated in observational studies that lacked an intervention or invasive procedure.
17. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
18. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within the past 2 years.
19. Is taking or expected to take an excluded medication.
20. Works a night (third) shift (defined as 11 PM [2300] to 7 AM [0700]). (Only for participants with ambulatory blood pressure monitoring [ABPM].)
21. Has an upper arm circumference <24 cm or >42 cm. (Only for participants with ABPM.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (30):
- China (30):
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tong Ren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi Zhuang
  - Affiliated Hospital of Hainan Medical University., Haikou, Hainan
  - Hebei Cangzhou Central Hospital, Cangzhou, Hebei
  - The 4th Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Hunan Province People's Hospital, Changsha, Hunan
  - Zhuzhou Central Hospital, Fuzhou, Hunan
  - Cardiology/Zhong Da Hospital, Southeast University, Nanjing, Jiangsu
  - Nanjing Medical University Affiliated 2nd Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Cardiology/The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Wu J, Du X, Lv Q, Li Z, Zheng Z, Xia Y, Tang C, Yao Z, Zhang J, Long M, Hisada M, Wu J, Zhou W, Ma C. A phase 3 double-blind randomized (CONSORT-compliant) study of azilsartan medoxomil compared to valsartan in Chinese patients with essential hypertension. Medicine (Baltimore). 2020 Aug 7;99(32):e21465. doi: 10.1097/MD.0000000000021465. PMID 32769878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in China from 27 August 2015 to 13 October 2017.
Pre-assignment Details: Participants with a diagnosis of hypertension were randomized at a ratio of 1:1:1 into 1 of 3 treatment groups, once a day azilsartan medoxomil 40 mg, azilsartan medoxomil 80 mg or valsartan 160 mg.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Started | 199 | 209 | 204
Completed | 189 | 189 | 183
Not Completed | 10 | 20 | 21
Not completed — Pretreatment Event/Adverse Event | 3 | 6 | 3
Not completed — Major Protocol Deviation | 1 | 4 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Voluntary Withdrawal | 6 | 5 | 10
Not completed — Lack of Efficacy | 0 | 3 | 3
Not completed — Reason not Specified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg | Total
Number analyzed (Participants) | 199 | 209 | 204 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.52) | 57.0 (9.88) | 56.8 (9.48) | 57.1 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 94 | 74 | 260
  Male | 107 | 115 | 130 | 352
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 199 | 209 | 204 | 612
Region of Enrollment [Count of Participants; unit: Participants]
  China | 199 | 209 | 204 | 612
Height [Mean (Standard Deviation); unit: cm] | 164.3 (8.92) | 164.2 (8.81) | 165.3 (7.73) | 164.6 (8.50)
Weight [Mean (Standard Deviation); unit: kg] | 71.75 (14.046) | 71.60 (11.903) | 72.79 (12.903) | 72.05 (12.952)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=(baseline weight in kg)/(height in cm)/100)^2
  kg/m^2 | 26.43 (3.784) | 26.47 (3.436) | 26.52 (3.444) | 26.48 (3.550)
Smoking Classification [Count of Participants; unit: Participants]
  Participant has never smoked | 151 | 147 | 136 | 434
  Participant is a current smoker | 39 | 51 | 55 | 145
  Participant is an ex-smoker | 9 | 11 | 13 | 33
Female Reproductive Status [Count of Participants; unit: Participants]
  Postmenopausal | 68 | 71 | 51 | 190
  Surgically Sterile | 12 | 5 | 7 | 24
  Female of Childbearing Potential | 12 | 18 | 16 | 46
  N/A (Participant is Male) | 107 | 115 | 130 | 352
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Calculated using the Modification of Diet in Renal Disease (MDRD) formula.
  mL/min/1.73m^2 | 109.50 (26.309) | 110.45 (28.771) | 108.00 (29.206) | 109.32 (28.116)
Baseline glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin] | 5.67 (0.569) | 5.77 (0.793) | 5.75 (0.716) | 5.73 (0.701)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Sitting Clinic Systolic Blood Pressure (SBP)
Description: The change in trough clinic sitting SBP measured at Week 8 relative to baseline. The trough is the average of the non-missing values of 3 serial trough sitting SBP measurements. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 8 blood pressure was measured approximately 24 hours after the previous day's dose.
Time Frame: Baseline and Week 8
Population: Full Analysis Set (FAS) included all randomly assigned participants who received at least 1 dose of double-blind study drug. Missing values were imputed using last observation carried forward (LOCF). Number analyzed at a visit is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
mm Hg
  Baseline SBP: number analyzed (Participants) | 197 | 206 | 197
  Baseline SBP | 157.873 (0.5123) | 158.236 (0.5010) | 158.594 (0.5123)
  Change at Week 8: number analyzed (Participants) | 197 | 206 | 197
  Change at Week 8 | -22.483 (1.0258) | -24.236 (1.0027) | -20.551 (1.0258)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Non-Inferiority — A test for noninferiority was done using a margin of 1.5 mm Hg. A test for significant difference was performed at 5% level; p = 0.184, ANCOVA — Change at Week 8: P-value was calculated using analysis of covariance (ANCOVA) model, with treatment group as a fixed effect and baseline trough sitting clinic SBP as a continuous covariate; Least Square Mean Difference = -1.932, 95% CI 2-sided [-4.782 to 0.918], Standard Error of Mean 1.4512
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.010, ANCOVA — Change at Week 8: P-value was calculated using ANCOVA model, with treatment group as a fixed effect and baseline trough sitting clinic SBP as a continuous covariate; Least Square Mean Difference = -3.685, 95% CI 2-sided [-6.502 to -0.868], Standard Error of Mean 1.4344

2. Secondary Outcome: Change From Baseline in Trough Sitting Clinic Diastolic Blood Pressure (DBP)
Description: The change in trough clinic sitting DBP measured at Week 8 relative to baseline. The trough is the average of the non-missing values of 3 serial trough sitting DBP measurements. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 8 blood pressure was measured approximately 24 hours after the previous day's dose.
Time Frame: Baseline and Week 8
Population: FAS included all randomly assigned participants who received at least 1 dose of double-blind study drug. Missing values were imputed using LOCF. Number analyzed at a visit is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
mm Hg
  Baseline DBP: number analyzed (Participants) | 197 | 206 | 197
  Baseline DBP | 91.790 (0.7306) | 91.510 (0.7145) | 92.298 (0.7306)
  Change at Week 8: number analyzed (Participants) | 197 | 206 | 197
  Change at Week 8 | -10.101 (0.6684) | -11.463 (0.6538) | -8.641 (0.6686)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.123, ANCOVA — Change at Week 8: P-value was calculated using ANCOVA model, with treatment group as a fixed effect and baseline trough sitting clinic DBP as a continuous covariate; Least Square Mean Difference = -1.459, 95% CI 2-sided [-3.316 to 0.397], Standard Error of Mean 0.9455
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.003, ANCOVA — Change at 8 Week: P-value was calculated using ANCOVA model, with treatment group as a fixed effect and baseline trough sitting clinic DBP as a continuous covariate; Least Square Mean Difference = -2.822, 95% CI 2-sided [-4.659 to -0.985], Standard Error of Mean 0.9354

3. Secondary Outcome: Percentage of Participants Who Achieved a Clinic SBP Response at Week 8
Description: Clinic SBP response was defined as clinic SBP <140 mm Hg and/or reduction of ≥20 mm Hg from Baseline. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 8 blood pressure was measured approximately 24 hours after the previous day's dose.
Time Frame: Week 8
Population: FAS included all randomly assigned participants who received at least 1 dose of double-blind study drug. Missing values were imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
percentage of participants | 67.0 | 68.9 | 69.0
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.548, Regression, Logistic — P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough SBP as a continuous covariate; Odds Ratio (OR) = 0.877, 95% CI 2-sided [0.571 to 1.347], Standard Error of Mean 0.1920
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.921, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.979, 95% CI 2-sided [0.638 to 1.501], Standard Error of Mean 0.2136

4. Secondary Outcome: Percentage of Participants Who Achieved a Clinic DBP Response at Week 8
Description: Clinic DBP response was defined as clinic DBP <90 mm Hg and/or reduction of ≥10 mm Hg from Baseline. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 8 blood pressure was measured approximately 24 hours after the previous day's dose.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
percentage of participants | 81.2 | 81.6 | 79.7
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.904, Regression, Logistic — P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough DBP as a continuous covariate; Odds Ratio (OR) = 1.033, 95% CI 2-sided [0.607 to 1.759], Standard Error of Mean 0.2805
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.790, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.074, 95% CI 2-sided [0.633 to 1.823], Standard Error of Mean 0.2897

5. Secondary Outcome: Percentage of Participants Who Achieved Both Clinic SBP and DBP Response at Week 8
Description: Clinic SBP response was defined as clinic SBP <140 mm Hg and/or reduction of ≥20 mm Hg from Baseline and clinic DBP response was defined as clinic DBP <90 mm Hg and/or reduction of ≥10 mm Hg from Baseline. Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 8 blood pressure was measured approximately 24 hours after the previous day's dose.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
percentage of participants | 62.9 | 67.0 | 64.5
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.624, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.901, 95% CI 2-sided [0.594 to 1.367], Standard Error of Mean 0.1916
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.647, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.103, 95% CI 2-sided [0.726 to 1.674], Standard Error of Mean 0.2350

6. Secondary Outcome: Percentage of Participants Who Achieved Target Clinic SBP <140 mm Hg, Clinic DBP <90 mm Hg or Both at Week 8
Description: Blood pressure was measured using a validated, automated device after the participant had been sitting for at least 5 minutes. Week 8 blood pressure was measured approximately 24 hours after the previous day's dose.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
percentage of participants
  Clinic SBP <140 mm Hg | 60.9 | 62.6 | 62.9
  Clinic DBP <90 mm Hg | 77.2 | 76.7 | 74.6
  Clinic SBP <140 mm Hg and DBP <90 mm Hg | 58.4 | 60.2 | 55.8
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.404, Regression, Logistic — Clinic SBP <140 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough SBP as a continuous covariate; Odds Ratio (OR) = 0.831, 95% CI 2-sided [0.537 to 1.284], Standard Error of Mean 0.1846
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.768, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.937, 95% CI 2-sided [0.606 to 1.447], Standard Error of Mean 0.2078
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.852, Regression, Logistic — Clinic DBP <90 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough DBP as a continuous covariate; Odds Ratio (OR) = 1.051, 95% CI 2-sided [0.620 to 1.784], Standard Error of Mean 0.2837
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.868, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; Odds Ratio (OR) = 1.045, 95% CI 2-sided [0.620 to 1.763], Standard Error of Mean 0.2788
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.847, Regression, Logistic — Clinic SBP<140 mm Hg and DBP<90 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough SBP as a continuous covariate; Odds Ratio (OR) = 1.042, 95% CI 2-sided [0.684 to 1.590], Standard Error of Mean 0.2244
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.460, Regression, Logistic — [p-value comment as in outcome 6, analysis 5]; Odds Ratio (OR) = 1.172, 95% CI 2-sided [0.769 to 1.785], Standard Error of Mean 0.2517

7. Secondary Outcome: Percentage of Participants Who Achieved Target Clinic SBP <130 mm Hg, Target Clinic DBP <80 mm Hg or Both at Week 8
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 199 | 209 | 204
percentage of participants
  Clinic SBP <130 mm Hg | 37.6 | 42.7 | 28.4
  Clinic DBP <80 mm Hg | 45.2 | 51.9 | 37.1
  Clinic SBP <130 mm Hg and DBP <80 mm Hg | 28.9 | 33.0 | 21.8
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.077, Regression, Logistic — Clinic SBP<130 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough SBP as a continuous covariate; Odds Ratio (OR) = 1.487, 95% CI 2-sided [0.958 to 2.307], Standard Error of Mean 0.3333
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.003, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.914, 95% CI 2-sided [1.241 to 2.951], Standard Error of Mean 0.4229
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.137, Regression, Logistic — Clinic DBP<80 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough DBP as a continuous covariate; Odds Ratio (OR) = 1.427, 95% CI 2-sided [0.893 to 2.280], Standard Error of Mean 0.3414
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.003, Regression, Logistic — Clinic DBP <80 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough DBP as a continuous covariate; Odds Ratio (OR) = 2.017, 95% CI 2-sided [1.263 to 3.220], Standard Error of Mean 0.4816
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg vs Valsartan 160 mg; Test type: Other; p = 0.140, Regression, Logistic — Clinic SBP<130 mm Hg and DBP<80 mm Hg: P-value was calculated using logistic regression model with treatment group as a fixed effect and baseline trough SBP as a continuous covariate; Odds Ratio (OR) = 1.424, 95% CI 2-sided [0.891 to 2.276], Standard Error of Mean 0.3407
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg vs Valsartan 160 mg; Test type: Other; p = 0.015, Regression, Logistic — [p-value comment as in outcome 7, analysis 5]; Odds Ratio (OR) = 1.769, 95% CI 2-sided [1.118 to 2.797], Standard Error of Mean 0.4136

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 14 days after the last dose of study drug (Up to Week 12)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg | Azilsartan Medoxomil 80 mg | Valsartan 160 mg
All-Cause Mortality (participants affected / at risk) | 1/199 | 0/209 | 0/204
Serious Adverse Events (participants affected / at risk) | 2/199 | 7/209 | 6/204
Other Adverse Events (participants affected / at risk) | 34/199 | 37/209 | 35/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg (N=199) | Azilsartan Medoxomil 80 mg (N=209) | Valsartan 160 mg (N=204)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Urate nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Ureteral cyst (Renal and urinary disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg (N=199) | Azilsartan Medoxomil 80 mg (N=209) | Valsartan 160 mg (N=204)
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 | 14 | 16
Upper respiratory tract infection (Infections and infestations) | 10 | 13 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 11 | 8
Albuminuria (Renal and urinary disorders) | 11 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02480764/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT02480764/SAP_001.pdf